CLINICAL TRIAL: NCT03580512
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Study to Evaluate the Feasibility of Integrating the Point-of-care Testing for Sexually Transmitted Infections and HIV Into Community-based Clinics for MSM and TGW in Thailand
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: POC HIV&STI
Record Dates: First submitted 2018-05-31; First posted 2018-07-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Men Who Have Sex With Men and Transgender Women
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Group 1: - 800 existing clients who already received PrEP
- Group 2: * 800 new clients who present for HIV testing and are HIV-negative. All will be offered PrEP
  * 600 clients who will refuse PrEP
  * 200 clients who will receive PrEP
- Group 3: - 400 new clients who are HIV-positive or new clients who present for HIV testing and are HIV-positive

SUMMARY:
This will be a prospective study that will enroll up to 2000 MSM and TG from community-based clinics in Bangkok, Chonburi, Chiang Mai, and Songkhla.

DETAILED DESCRIPTION:
Eligible participants will be followed up until the completion of a 12-month period. All participants will be followed up every 3 months. An additional follow up visit at month 1 will be made for participants who PrEP is initiated at entry visit (those who already received PrEP prior to the study will not need the additional visit).

Study Sites

The study will take place at the following community-based clinics:

1. SWING DIC, Bangkok, Thailand
2. RSAT DIC, Bangkok, Thailand
3. SWING DIC, Chonburi, Thailand
4. Sisters DIC, Chonburi, Thailand
5. Mplus DIC, Chiang Mai, Thailand
6. RSAT DIC, Songkhla, Thailand

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Age ≥ 18 years old
3. Men or transgender women who have sex with men
4. Have at least one of the following risks for HIV acquisition in the past 6 months:

   * Any unprotected receptive anal sex
   * More than 5 sexual partners, regardless of condom use and serostatus
   * History of syphilis, chlamydia or gonorrhea diagnosed or treated
   * Any stimulant drug use
5. Have signed the consent form

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Approximately 2000 MSM and TG
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who receive same-day diagnosis and treatment of CT/NG in community-based clinics | 1 years
Proportion of participants who receive same-day diagnosis of HIV infection in community-based clinics | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Nittaya Phanuphak, MD, PhD, Principal Investigator — Thai Red Cross AIDS Research Centre (TRCARC)
Locations (6):
- Thailand (6):
  - 1.Swing Dic,, Bangkok
  - 2.Rsat Dic,, Bangkok
  - 5. Mplus DIC,, Chiang Mai
  - 3.Swing Dic, Chon Buri
  - 4. Sisters DIC,, Chon Buri
  - 6.Rsat Dic,, Songkhla

REFERENCES:
- [Derived] Hiransuthikul A, Sungsing T, Jantarapakde J, Trachunthong D, Mills S, Vannakit R, Phanuphak P, Phanuphak N. Correlations of chlamydia and gonorrhoea among pharyngeal, rectal and urethral sites among Thai men who have sex with men: multicentre community-led test and treat cohort in Thailand. BMJ Open. 2019 Jun 27;9(6):e028162. doi: 10.1136/bmjopen-2018-028162. PMID 31253622
- [Derived] Hiransuthikul A, Janamnuaysook R, Sungsing T, Jantarapakde J, Trachunthong D, Mills S, Vannakit R, Phanuphak P, Phanuphak N. High burden of chlamydia and gonorrhoea in pharyngeal, rectal and urethral sites among Thai transgender women: implications for anatomical site selection for the screening of STI. Sex Transm Infect. 2019 Nov;95(7):534-539. doi: 10.1136/sextrans-2018-053835. Epub 2019 Apr 13. PMID 30982000